CLINICAL TRIAL: NCT05123755
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2a Multiple Ascending Dose Study to Examine the Safety, Tolerability and Efficacy of AV-001 Injection in Patients Hospitalized With Pneumonia Due To COVID-19 or Other Respiratory Infections.
Brief Title: Phase 2a Multiple Ascending Dose Study in Hospitalized Patients With Pneumonia.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vasomune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV001-004; CDMRP-PR203503 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2021-11-08; First posted 2021-11-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Respiratory Distress Syndrome; Viral or Bacterial Infections; Pneumonia; Pneumonia, Viral; Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Bacterial Infections; Pneumonia; Pneumonia, Viral; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: This is a randomized (1:1 ratio) placebo controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, placebo-controlled study. All sponsor, vendor and site study staff will be blinded to treatment assignment, with the exception of the unblinded biostatistician, unblinded site pharmacist, and unblinded site monitor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AV-001 Injection with standard of care (SOC). (Active Comparator): A total of 120 eligible patients (20 patients in each of cohort 1, 2 and 3 and 60 patients in cohort 4) will be randomized in a 1:1 ratio to receive either AV-001 Injection or AV-001 placebo Injection, together with standard of care (SOC). Doses of AV-001 Injection will start with 12.5 μg/kg/day in cohort 1 and are anticipated to increase to 25 μg/kg/day in cohort 2, 56 μg/kg/day in cohort 3 and to be determined (TBD) in cohort 4. The dose for cohort 4 will be determined by the Data Safety Monitoring Board (DSMB) based on emerging data from cohorts 1, 2 and 3.
  Interventions: Drug: AV-001 Injection
- AV-001 Placebo Injection with standard of care (SOC). (Placebo Comparator): A total of 120 eligible patients (20 patients in each of cohort 1, 2 and 3 and 60 patients in cohort 4) will be randomized in a 1:1 ratio to receive either AV-001 Injection or AV-001 placebo Injection, together with standard of care (SOC).
  Interventions: Drug: AV-001 Placebo Injection

INTERVENTIONS:
Drug: AV-001 Injection — AV-001 (mpaBr) Cl for Injection 2.5 mg/mL
  Arms: AV-001 Injection with standard of care (SOC).
Drug: AV-001 Placebo Injection — D-PBS
  Arms: AV-001 Placebo Injection with standard of care (SOC).

SUMMARY:
A Phase 2a, randomized, double-blind, placebo-controlled, multiple ascending dose study in patients who are hospitalized with presumed pneumonia requiring supplemental oxygen therapy. The purpose of this study is to examine the safety, tolerability and efficacy of AV-001 Injection administration daily to the earlier of day 28 or EOT (day prior to hospital discharge). A total of 120 eligible patients (20 patients in each of cohort 1, 2 and 3 and 60 patients in cohort 4) will be recruited from up to 25 participating institutions/hospitals. Patients will be randomized in a 1:1 ratio to receive either AV-001 Injection or AV-001 placebo Injection, together with standard of care (SOC).

DETAILED DESCRIPTION:
Pneumonia is a leading cause of hospitalization among adults and children in the United States and has ranked among the top 10 causes of death according to the CDC. A large variety of microorganisms can cause pneumonia including respiratory viruses, bacteria and fungi and there are great geographic variations in their prevalence. In the United States, common causes of viral pneumonia are SARS-CoV-2, influenza and respiratory syncytial virus (RSV) and bacterial pneumonia are Streptococcus pneumoniae (pneumococcus).

Emerging evidence indicates that the respiratory system mechanics of patients with typical ARDS, with or without COVID-19 are broadly similar in contrast to earlier reports that suggested COVID-19-associated ARDS has distinctive features. SOC for patients with ARDS remains limited with current interventions that focus primarily on supportive therapy, including fluid management strategies and further injury prevention via lung protective ventilation. Ventilation approaches remain the cornerstone in the treatment of ARDS and approaches to minimize ventilator-induced lung injury (VILI) resulting from the imposition of stretch-trauma to the lung, continue to be a major focus of clinical importance. Several techniques may be utilized to accomplish this objective. Clinical guidelines strongly recommend volume-limited or pressure-limited ventilator approaches for patients with severe ARDS and high positive-end expiratory pressure strategies for patients with moderate to severe ARDS. Despite decades of improving supportive care, mortality remains high, ranging from 34.9% of patients with mild ARDS to 46.1% of patients with severe ARDS.

Whatever the causative organism it is increasingly apparent that their impact on lung microvasculature is a major contributing factor to morbidity and mortality associated with those infections. Most deaths from influenza virus infections occur due to pulmonary complications, in particular the development of acute respiratory distress syndrome (ARDS), that is due to increased permeability of the lung microvasculature. Emerging evidence in COVID-19 infections suggest a similar pathophysiology where pulmonary endothelial cells and vascular dysfunction contribute to the initiation and propagation of ARDS by altering blood vessel integrity, promoting a pro-coagulative state, inducing endotheliitis and mediating inflammatory cell infiltration. Therefore, a therapeutic intervention that could modulate the course of pulmonary disease not by treating the causative organism but by reducing the deleterious inflammatory sequalae of those infections may have a significant positive impact

AV-001 is a synthetic Angiopoietin-1 (Angpt-1) mimetic that has been shown to activate the Tie2 receptor tyrosine kinase; a transmembrane protein target most highly expressed on the surface of endothelial cells in the vasculature. The Tie2/Angiopoietin signaling axis has been identified as a nonredundant gatekeeper of vascular homeostasis. In healthy individuals, Tie2 is highly activated and signals the endothelium to fortify intracellular junctions and reduce expression of adhesion molecules, which serve as leukocyte tethers upon inflammation. As such, homeostatic activation results in the promotion of barrier defense against vascular leakage.

A total of 120 eligible patients (20 patients each in cohorts 1, 2 and 3 and 60 patients in cohort 4) will be recruited from participating institutions / hospitals. Patients will be randomized in a 1:1 ratio to receive either AV-001 Injection or AV-001 placebo Injection, together with SOC. All patients will receive supportive care according to the SOC for the trial site hospital likely to include remdesivir and or dexamethasone. Study drug will be administered by bolus IV injection (< 60 seconds). Doses of AV-001 Injection to be administered will start with the lowest proposed dose of 12.5 μg/kg/day in cohort 1 (DL1) and are anticipated to increase to 25 μg/kg/day in cohort 2 (DL2), 56 μg/kg/day in cohort 3 (DL3) and to be determined (TBD) based on recommendation from the DSMB for cohort 4 (DL4). The dose for cohort 4 will be chosen based on available safety and efficacy data obtained from all patients completing DL1, DL2 and DL3. DL4 may be an intermediate dose level, repeat of an earlier dose level (DL1, DL2, or DL3) or expansion of earlier dose level cohort (DL1, DL2, or DL3). Based on emerging data, a decision to enroll a fifth cohort (n=20 to increase the sample size to n=140) may also be made for the purpose of investigating an intermediate dose level, evaluating effects in patients with a different baseline Clinical Progression Scale (CPS) score or to provide comparative data regarding AV-001 Injection in patients with other respiratory viruses.

The study population for this Phase 2a study will consist of male and non-pregnant female patients, ≥ 18 years of age, hospitalized with presumed pneumonia secondary to SARS-CoV-2 or other viral or bacterial infection with acute onset to a respiratory compromise requiring supplemental oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give signed informed consent
* Patients hospitalized with a presumed diagnosis of pneumonia of < 48 hours duration requiring supplemental oxygen therapy. Eligible patients include those hospitalized for a separate non-infectious reason who subsequently develop a presumed pneumonia;
* Radiologic imaging (chest x-ray, CT scan, etc.) evidence of pulmonary involvement with new and persistent or progressive and persistent infiltrate, consolidation or cavitation.

Signs and symptoms:

At least 1 of the following signs:

* respiratory rate > 30 breaths/min;
* fever (> 38.0ºC or > 100.4o F);
* leukopenia (≤ 4,000 WBC/mm3 or leukocytosis (≥ 12,000 WBC/mm3);
* adults ≥ 70 years of age; altered mental status with no other recognized cause;

AND at least 1 of the following symptoms:

* New onset of purulent sputum or change in character of sputum or increased respiratory secretions;
* New onset or worsening cough, or dyspnea, or tachypnea;
* Rales or bronchial breath sounds;

  * Female patients of reproductive potential must be on an effective contraceptive method

Exclusion Criteria:

* Pregnant and/or lactating women
* Patients included in any other interventional trial
* Use of endotracheal intubation and mechanical ventilation or extracorporeal membrane oxygenation (ECMO) at screening
* Any concurrent serious medical condition or concomitant medication that would preclude participation in the study including but not limited to:

  * Septic shock as defined by systolic blood pressure (SBP) < 90 mmHg or diastolic blood pressure (DBP) of < 60 mmHg;
  * Multiple organ failure;
  * Are moribund irrespective of the provision of treatments;
  * Any significant bleeding disorder or vasculitis;
  * Any serious, nonhealing wound, peptic ulcer or bone fracture;
  * Liver cirrhosis;
  * History of a hypertensive crisis or hypertensive encephalopathy, or current, poorly controlled hypertension or hypotension;
  * Severe renal insufficiency or end stage renal disease as determined by estimated glomerular filtration rate <30mL/min/1.73m2;
  * ARDS risk factors of aspiration pneumonia, non-cardiac shock, trauma, blood transfusion or drug overdose.
* Any thromboembolic event within the past 3 months;
* Symptomatic congestive heart failure or symptomatic or poorly controlled cardiac arrhythmia > class II as per New York Heart Association (NYHA) classification;
* History of autonomic disorders or uncontrolled hypotension
* Hypersensitivity to drug products containing polyethylene glycol (PEG)
* Any other condition which the Principal Investigator feels may jeopardize the safety of the patient or the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of multiple doses of IV administrations of AV-001 Injection compared with AV-001 placebo Injection in hospitalized patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 60
  * Number of patients with any serious adverse event (SAE) (day 1 to 60/EOS)
  * Number of patients with any treatment emergent adverse event (TEAE) (day 1 to 60/EOS) AE assessments (day 1 to 60/EOS)

SECONDARY OUTCOMES:
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Measured as proportion of patients achieving a 2-point improvement in WHO COVID-19 CPS score from baseline and alive by day 28.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Time to first 2-point WHO CPS improvement using a Kaplan-Meier lifetable
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Measured as survival at day 28, displayed with a Kaplan- Meier lifetable.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Measured as proportion of patients that progress to respiratory failure by day 28.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Measured as proportion of patients that progress to mechanical ventilation by day 28.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Measured as proportion of patients with disease improvement of at least 1 point on the WHO COVID-19 CPS for 3 consecutive days and sustained the improvement through day 28.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  SpO2 saturation (up to day 28): measured as proportion of patients achieving normalization (last oxygen saturation of arterial blood [SaO2] value > 95%).
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Oxygen delivery: measured as the product of flow rate and volume per day.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Measured as the acute kidney injury stage distribution over time using the Kidney Disease Improving Global Outcomes (KDIGO) definition of Acute Kidney Injury (AKI).
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Measured as proportion of patients alive and discharged from the intensive care unit (ICU) at day 28.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Measured as proportion of patients alive and discharged from hospital at day 28.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 28
  Measured as time to hospital discharge status (discharge or day 28, whichever is earlier).

OTHER OUTCOMES:
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 60
  Measured as alive at day 60, displayed with a Kaplan- Meier lifetable.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 14
  Measured as proportion of patients that progress to respiratory failure by day 14.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 14
  Measured as proportion of patients that progress to mechanical ventilation by day 14.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 14
  Proportion of patients achieving a 2-point improvement in WHO COVID-19 CPS score from baseline and alive by day 14.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 14
  Measured as proportion of patients alive and discharged from the intensive care unit (ICU) at day 14.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 14
  Measured as proportion of patients alive and discharged from hospital at day 14.
Efficacy of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection in patients hospitalized with pneumonia due to COVID-19 and/or other respiratory infections | Up to Day 60
  Measured as durable loss of eGFR (by day 28 and day 60) from baseline (89-60 mL/min, 59-45 mL/min, 30-44 mL/min, <30 mL/min) or the development of severe AKI requiring continuous renal replacement therapy (CRRT), prolonged intermittent renal replacement therapy (PIRRT) or hemodialysis.
Effect of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection on exploratory biomarkers of Tie2 target engagement | Up to Day 28
  Measured as ratio of phosphorylated Tie2/Total Tie2 using flow cytometry analysis.
Effect of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection on exploratory biomarkers (Angpt-1, Angpt-2, and circulating Tie2). | Up to Day 28
  Measured using quantitative ELISA.
Effect of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection on disease biomarkers IL-6 in patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Measured at screening and at pre-dose on days 2, 4, 7, 10, 13, 16, 19, 22, 25 and the earlier of day 28 or EOT using quantitative reverse transcriptase polymerase chain reaction (RT-PCR) assay.
Effect of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection on disease biomarker IL-8 in patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Measured at screening and at pre-dose on days 2, 4, 7, 10, 13, 16, 19, 22, 25 and the earlier of day 28 or EOT using quantitative reverse transcriptase polymerase chain reaction (RT-PCR) assay.
Effect of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection on disease biomarkers TNFr-1 in patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Measured at screening and at pre-dose on days 2, 4, 7, 10, 13, 16, 19, 22, 25 and the earlier of day 28 or EOT using quantitative reverse transcriptase polymerase chain reaction (RT-PCR) assay.
Effect of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection on disease biomarker MCP-1 in patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Measured at screening and at pre-dose on days 2, 4, 7, 10, 13, 16, 19, 22, 25 and the earlier of day 28 or EOT using quantitative reverse transcriptase polymerase chain reaction (RT-PCR) assay.
Effect of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection on disease biomarker IP-10 in patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Measured at screening and at pre-dose on days 2, 4, 7, 10, 13, 16, 19, 22, 25 and the earlier of day 28 or EOT using quantitative reverse transcriptase polymerase chain reaction (RT-PCR) assay.
Effect of multiple IV administrations of AV-001 Injection compared with AV-001 placebo Injection on disease biomarker ICAM-1, in in patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Measured at screening and at pre-dose on days 2, 4, 7, 10, 13, 16, 19, 22, 25 and the earlier of day 28 or EOT using quantitative reverse transcriptase polymerase chain reaction (RT-PCR) assay.
PK as measured by Cmax of AV-001 Injection in hospitalized patients with severe COVID-19 disease. | Up to Day 28
  Assessment of the PK of AV-001 Injection in hospitalized patients with severe COVID-19 disease using population PK for DL1, DL2 and DL3. PK measured as Cmax from sample timepoints Pre-dose, 5 min, 30 min, 1, 2, 4, and 24 hours post-dose on days 1, 7 and the earlier of day 28 or EOT.
PK as measured by Tmax of AV-001 Injection in hospitalized patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Assessment of the PK of AV-001 Injection in hospitalized patients with pneumonia due to COVID-19 and/or other respiratory infections using population PK for DL1, DL2 and DL3. PK measured as Tmax, from sample timepoints Pre-dose, 5 min, 30 min, 1, 2, 4, and 24 hours post-dose on days 1, 7 and the earlier of day 28 or EOT.
PK as measured by AUC of AV-001 Injection in hospitalized patients with pneumonia due to COVID-19 and/or other respiratory infections. | Up to Day 28
  Assessment of the PK of AV-001 Injection in hospitalized patients with pneumonia due to COVID-19 and/or other respiratory infections using population PK for DL1, DL2 and DL3. PK measured as AUC from sample timepoints Pre-dose, 5 min, 30 min, 1, 2, 4, and 24 hours post-dose on days 1, 7 and the earlier of day 28 or EOT.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Denver Health Medical Center, Denver, Colorado
  - University of Florida College of Medicine, Jacksonville, Jacksonville, Florida
  - MedStar Health Research Institute, Inc., Hyattsville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No